CLINICAL TRIAL: NCT01832285
Title: Effect of Fluvoxamine Augmentation on Cognitive Function , Aggressive Behavior , Clinical Symptoms and mRNA and Protein Expression in Human Peripheral Mononuclear Blood Cells (PMC) in Medicated Schizophrenia Patients
Brief Title: Effect of Fluvoxamine on Cognition, Behavior, Symptoms and mRNA and Protein Expression in Schizophrenia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120241
Record Dates: First submitted 2013-02-14; First posted 2013-04-16 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-01

CONDITIONS: SCHIZOPHRENIA 1 (Disorder)
Keywords: fluvoxamine; cognition; schizophrenia; protein expression
MeSH Terms: conditions — Schizophrenia | interventions — Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluvoxamine (Experimental): Tablets of Fluvoxamine in dosage 100mg/day will be added to the treatment regimen and continued for 6 weeks
  Interventions: Drug: fluvoxamine

INTERVENTIONS:
Drug: fluvoxamine — 100mg/day, PO(in the mouth) each day during 6 weeks
  Other Names: Favoxile

SUMMARY:
The purpose of this study is to determine effect of Fluvoxamine augmentation on cognitive function , aggressive behavior , clinical symptoms and mRNA (messenger ribonucleic acid) and protein expression in human peripheral mononuclear blood cells (PMC) in medicated schizophrenia patients

DETAILED DESCRIPTION:
Clinical studies have shown that adding selective serotonin reuptake inhibitor (SSRI) antidepressants to antipsychotics can improve negative symptoms of schizophrenia in patients unresponsive to antipsychotics alone . The effect of SSRI augmentation on cognitive impairments of the illness which do not respond to antipsychotics and are associated with poor outcome has not been adequately tested .

In a recent study we showed that SSRI augmentation alters expression of gamma-aminobutyric acid(GABA A) receptor, protein kinase(PKC), brain-derived neurotrophic factor(BDNF) and related systems in peripheral mononuclear blood cells (PMC)of schizophrenia patients . There is evidence that these systems are abnormal in schizophrenia patients and are associated with cognitive and negative symptoms strengthening the likelihood that their modulation by SSRI augmentation can improve cognitive impairments .

Behavioral disturbance , particularly aggression is another feature of schizophrenia which is difficult to treat and leads to social and legal complications and poor outcome. Aggression is associated with serotoninergic dysfunction and there is evidence that SSRI can modify aggressive behavior including in schizophrenia patients .Thus this study will also examine the effect of SSRI augmentation on aggressive behavior and other behavioral and functional measures .

The mechanism of SSRI augmentation is not known and is the focus of research interest.

We have recently shown in laboratory studies that combined treatment of SSRI antidepressant and antipsychotic drug resulted in biochemical changes, different from the effects of the individual medications. Changes unique to the combined treatment were found in GABAergic components and related systems including GABA-Aβ3 receptor, glutamic acid decarboxylase 67 and PKCβ in selected areas of rat brain and in cultures of cortical neurons. Studies of drug mechanisms in humans have utilized blood products and PMC which are readily accessible and may reflect molecular processes in the central nervous system (CNS) of schizophrenic patients .Using this method in schizophrenia patients treated with SSRI augmentation we showed that changes in mRNA encoding for GABA A receptor , PKC and related proteins were associated with clinical improvement indicating that the changes observe in the laboratory have clinical relevance.

Methods The dose of antipsychotics will be unchanged for at least 2 weeks prior to the study and will remain steady throughout the study period. Fluvoxamine 100mg/day will be added to the treatment regimen and continued for 6 weeks. Clinical state will be assessed using validated rating scales and cognitive performance will be assessed with a cognitive test battery. Behavior and function , including s will be assessed with appropriate scales Blood samples will be taken at baseline and at 1, 3 and 6 weeks.At the end of the study protocol (after 6 weeks) the patients will be given the option to continue receiving the fluvoxamine. It can be assumed that the included subjects would not have received fluvoxamine if it weren't for their participation in the study for lack of indication for their primary diagnosis (see inclusion criteria below). The PMC's will be assayed using microarray, (PCR) polymerase chain reaction and proteomic techniques. Changes in RNA and protein expression will be detected and compared with changes in clinical symptoms , cognitive function and behavioral change . Identification of biochemical changes related to augmentation treated and their relation to symptomatic and cognitive changes will be the major potential benefit of the study.

Subjects 40 chronic schizophrenic or schizoaffective patients (DSM-IVTR)who have persistent negative symptoms and cognitive impairment despite adequate treatment will participate. The sample will include patients with a history of aggressive behavior hospitalized in the forensic wards and as well as patients in regular hospital wards and outpatients settings.

Assessments The diagnosis will determined by a consensus of two senior psychiatrists using the DSM-IVTR criteria. Physical assessment (which includes a physical examination as well as measurements of blood pressure and pulse) will be taken from the patient's medical records prior to the commencement of the study. Background and demographic characteristics, details of the present illness, medications, general medical history and current laboratory tests will also be evaluated.

Clinical state and cognitive function will be assessed prior to fluvoxamine treatment and then during the study period according to the flow sheet below.

Clinical assessment scales will include:

Schedule for the Assessment of Negative Symptoms (SANS); Schedule for the Assessment of Positive Symptoms (SAPS); Simpson Angus Scale for Extrapyramidal Side Effects; Abnormal Involuntary Movement Scales (AIMS); Calgary Depression Scale

Cognitive assessment will include:

Mini Mental State Examination, Dot test, Digit Span, Finger Tap Test modified, Wechsler memory tests. Computerized Cognitive Neuropsychological Battery:Computerized judgment of line orientation (CJOLO); Penn face memory test (PFMT); Visual object learning test (VOLT); Abstraction inhibition and working memory task (AIM), Identification of facial emotions (PEAT); Differentiation of facial emotion (EMDIF).

Behavioral and function assessment Overt aggression Scale GAF (DSM IV TR) Critical Events Blood tests Approx 50cc of blood will be taken at baseline, prior to start of fluvoxamine treatment, and 1,3 and 6 weeks after the start of fluvoxamine treatment.

Treatment of blood samples: Blood will be collected into heparinized tubes, kept on ice and transported to the laboratory. Blood samples will be processed to enable assay of PMC elements of interest, including chemokine receptors, G protein receptors such as the GABAA receptor , their regulators such as, PKC GSK3 RGS7 and neurotrophins such as BDNF.

Some of the serum will be frozen for subsequent analyses of antipsychotic drug and neurohormone concentration. The blood samples will be stored in the molecular neuropsychiatry laboratory at the Technion Institute of Technology (Haifa) under the supervision of the principal investigator, Prof. Henry Silver. The samples will be unnamed and numbered. They will be kept for a maximum of 10 years. The participants will be given the option to ask for the destruction of the samples at any time.

Flow sheet Week 0 Subject entry Clinical assessment Cognitive Assessment Behavioral Assessment Blood collection- baseline Start Fluvoxamine Week 1 Blood collection Week 3 Clinical assessment Cognitive assessment Behavioral Assessment Blood collection Week 6 Clinical assessment Cognitive assessment Behavioral Assessment Blood collection

Implementation of the protocol The implementation of the protocol will involve a team of research clinicians from Sha'ar Menashe Mental Health Center (Hadera) as well as the Technion Institute of Technology (Haifa) under the direction of the principal investigator, Prof. Henry Silver. Clinical and cognitive ratings will be each respectively obtained by one rater in order to eliminate inter-rater bias.

Statistical analysis Statistical analysis of all studied parameters will be done between repeated measures using analysis of variance (ANOVA) and the t-test. For nonparametric distributions the Mann Whitney U test and the chi test will be utilized.

Risk/Benefit and Safety Considerations The taking of blood sample is the only invasive procedure. This is a routine procedure accompanied by minor discomfort. Fluvoxamine augmentation has been studied extensively and has been used safely in numerous studies. Side effects of fluvoxamine include nausea and GI disturbance. The side effects will be determined during the clinical assessments on weeks 0,3 and 6 according to the flow sheet above using a clinical interview as well as a physical examination when necessary. The side effects will be documented in the study protocol. Severe adverse events will be monitored by the treating physicians and reported to the team of research clinicians.

The major advance of this methodology is that it enables the detection of RNA and protein changes in PMC by assigning each subject as his/her own control, and will enable change in clinical state to be related to the biochemical changes. Thus, the direct potential benefit for the participants in this study would be improvement cognitive ,behavioral (including aggressive ) and clinical symptoms, consequently improving their potential for well being and rehabilitation while the major potential benefit for society would be the identification of molecular changes accompanying clinical response to SSRI augmentation as a basis for the understanding of their pharmacological mechanism of action and consequently opening new vistas for treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* A diagnosis of schizophrenia (DSM-IVTR)
* Antipsychotic dose unchanged for at least 2 weeks prior to study
* SANS score>= 3 on at least one of the global measures of affective blunting, alogia or avolition.
* Knowledge of Hebrew

Exclusion Criteria:

* Dementia or other serious neurological disorders
* History of alcohol or drug use
* Patients with a legal guardian
* Patients involuntarily hospitalized by order of the district psychiatrist
* Use of antidepressants within 1 month of the study
* Renal or hepatic disorder
* Patients with upper GI bleeds
* Patients with SIADH syndrome
* Pregnant woman

Criteria for the cessation of the study after initial commencement

* Severe adverse events (including but not only GI, cardiovascular, neurologic, hematologic or urologic severe adverse events)
* Emergent suicidality
* Emergence of hypomanic or manic symptoms
* If the subject requests to stop

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
effect of SSRI augmentation on cognitive function in schizophrenia patients | 1 year
  Clinical state and cognitive function will be assessed prior to fluvoxamine treatment and then during the study period according to the flow sheet below.
  Clinical assessment scales will include:Schedule for the Assessment of Negative Symptoms (SANS),Schedule for the Assessment of Positive Symptoms (SAPS) Simpson Angus Scale for Extrapyramidal Side Effects (SA); Abnormal Involuntary Movement Scales (AIMS); Calgary Depression Scale ,Cognitive assessment will include:Mini Mental State Examination, Dot test , Modified , Digit Span, Finger Tap Test, modified, Wechsler memory tests, Computerized Cognitive Neuropsychological Battery:Computerized judgment of line orientation (CJOLO); Penn face memory test (PFMT); Visual object learning test (VOLT); Abstraction inhibition and working memory task (AIM), Identification of facial emotions (PEAT); Differentiation of facial emotion (EMDIF).
  Behavioral and function assessment , Overt aggression Scale, GAF (DSM IV TR) Critical Events

SECONDARY OUTCOMES:
effect of SSRI augmentation on the RNA and protein products in peripheral mononuclear cells | 1 year
  Approx 50cc of blood will be taken at baseline,and 1,3 and 6 weeks after the start of fluvoxamine treatment.
  Blood will be collected into heparinized tubes, kept on ice and transported to the laboratory. Blood samples will be processed to enable assay of PMC elements of interest, including chemokine receptors, G protein receptors such as the GABAA receptor , their regulators such as, PKC GSK3 RGS7 and neurotrophins such as BDNF.
  Some of the serum will be frozen for subsequent analyses of antipsychotic drug and neurohormone concentration. The blood samples will be stored in the molecular neuropsychiatry laboratory at the Technion Institute of Technology (Haifa) under the supervision of the principal investigator, Prof. Henry Silver. The samples will be unnamed and numbered. They will be kept for a maximum of 10 years. The participants will be given the option to ask for the destruction of the samples at any time.

CONTACTS AND LOCATIONS:
Overall Officials: Silver Henry, Professor, Principal Investigator — Shaar Menashe Mental Health Center Affilated to Medical Faculty of Technion University
Locations (1):
- Shaar Menashe Mental Health Center, Hadera, Ha Sharon, Israel